CLINICAL TRIAL: NCT03451084
Title: A Phase IIA Dose Optimisation Study of ASLAN003 in Acute Myeloid Leukemia
Brief Title: A Dose Optimisation Study of ASLAN003 in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN003-003
Record Dates: First submitted 2018-01-23; First posted 2018-03-01 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML, ASLAN, DHODH
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Dose Level 1 (Experimental)
  Interventions: Drug: ASLAN003
- Part 1: Dose Level 2 (Experimental)
  Interventions: Drug: ASLAN003
- Part 1: Dose Level 3 (Experimental)
  Interventions: Drug: ASLAN003
- Part 1: Dose Level 4 (Experimental)
  Interventions: Drug: ASLAN003
- Part 2:ASLAN003 at Optinum Dose Level -1 & Azacitidine (Experimental)
  Interventions: Drug: ASLAN003
- Part 2:ASLAN003 at Optinum Dose Level & Azacitidine (Experimental)
  Interventions: Drug: ASLAN003

INTERVENTIONS:
Drug: ASLAN003 — Patients will be administered with the study drug, ASLAN003. The study drug is to be administered orally, QD or BID. It is recommended to administer the study drug with food or within 30 minutes after food intake.

SUMMARY:
ASLAN003-003 is a multi-center, Phase IIA study to evalute the efficacy of ASLAN003 in AML patients who are ineligible for standard treatment with an expansion cohort in relapsed/refractory patients, and to determine the appropriate dose of ASLAN003 in combination with azacitidine in older (more than or equal to 60 years) AML patients who have exhausted any approved and available treatment options.

DETAILED DESCRIPTION:
ASLAN003-003 is a multi-center, Phase IIA study to determine the optimum dose of ASLAN003 based on the safety, efficacy, and tolerability of varying doses of ASLAN003 (100 mg QD, 200 mg QD, 100 mg BID, and possibly 200 mg BID) administered to AML subjects daily for a continuous 28-day treatment cycle until disease relapse, disease progression, unacceptable toxicity, or withdrawal of consent.

The study has 2 parts and plans to enroll a total of 44 to 56 patients with 18 to 24 patients in Part 1 and 26 to 32 patients in Part 2 (comprising Parts 2A and 2B). The Overall Complete Remission Rate will be evaluated in AML patients not eligible for standard treatment (Part 1) and in relapsed and refractory AML patients (Part 2A) using the optimum dose of ASLAN003 established in Part 1 of the study. In Part 2B of the study, the appropriate dose of ASLAN003 in combination with azacitidine in older (more than or equal to 60 years) AML patients who have exhausted any approved and available treatment options will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are of or older than 18 years old in the United States or are of or older than the legal age in the respective countries at the time when written informed consent is obtained
2. Patients who are able to understand and willing to sign the informed consent form (ICF)
3. Patients who are diagnosed with AML according to the 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia (refer to Appendix 1: WHO Classification of Acute Myeloid Leukemia)
4. Patients who have a sufficient archival or fresh BM aspiration sample for the evaluation of relevant exploratory endpoint.

Note: Patients who do not have sufficient archival BM aspiration sample and refuse to repeat the procedure may be enrolled in the trial only after written confirmation by ASLAN 5. Part 1: Patients who are ineligible for standard treatment of AML including to the following conditions:

* Patients who are ineligible for chemotherapy, and have exhausted any approved and available treatment options. More details on patients who are considered as ineligible or unfit for chemotherapy as per Ferrara et al, Leukemia, 2013 can be found in Appendix 4.
* Patients who have relapsed from prior remission;
* Patients who have failed to respond to prior therapy including chemotherapy, hypomethylating agents, and bone marrow transplantation.

  5. Part 2A: Patients who have relapsed or refractory AML to treatments including chemotherapy, hypomethylating agents, bone marrow transplantation, and other anti-leukemic agents
  * Relapsed patients who have bone marrow blasts ≥5%; or reappearance of blasts in the blood; or development of extramedullary disease after prior CR or CRi
  * Refractory patients who have no CR or CRi after 2 courses of intensive induction treatment 5. Part 2B: Older patients (more than or equal to 60 years) AML patients who have exhausted any approved and available treatment options.

    6. Patients who have an ECOG performance status of ≤ 2 7. Patients with adequate renal and hepatic function, as defined below:
* Estimated Glomerular Filtration Rate (eGFR) or creatinine clearance (CrCl) (CrCl calculated by the Cockroft and Gault method) ≥ 40 ml/min/1.73 m2
* Total bilirubin, AST, and ALT ≤ 1.5 × ULN

Exclusion Criteria:

1. Patients who are diagnosed with de novo myeloid sarcoma without BM involvement
2. Patients who are diagnosed with acute promyelocytic leukemia/retinoic acid receptor alpha (PML-RARA)
3. Patients who received any other standard or investigational treatment for their leukemia within the last 7 days before starting the first dose of study drug, with the exception of leukapheresis and hydroxyurea
4. Patients with unresolved serious toxicity (≥ CTCAE 4.03 Grade 2) from prior administration of standard or investigational treatment for their leukemia
5. Patients who have a positive test for human immunodeficiency virus (HIV), viral hepatitis C infection (patients with sustained viral response are not excluded), active viral hepatitis B infection (positive hepatitis B surface antigen [HBsAg]) with hepatitis B virus deoxyribonucleic acid (DNA) exceeding 2000 IU/ml
6. Patients who have a known history of liver cirrhosis Child-Pugh score B or C
7. Patients who have any history of other malignancy unless in remission for more than 1 year (skin carcinoma and carcinoma-in-situ of uterine cervix treated with curative intent is not exclusionary)
8. Female patients who are pregnant or breast-feeding
9. Patients with a known history of alcohol or drug addiction on the basis that there could be a higher risk of non-compliance to study treatment
10. Patients with a history or presence of a clinically significant condition which in the opinion of the Investigator could jeopardize the safety of the patient or the validity of the study results
11. Patients who have been previously treated with ASLAN003

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- 1 Site, Louisville, Kentucky, United States
- Australia (6):
  - 1 Site, Albury, New South Wales
  - 3 Sites, Darlinghurst, New South Wales
  - 1 Site, Waratah, New South Wales
  - 1 Site, Douglas, Queensland
  - 1 Site, Adelaide, South Australia
  - 3 Sites, Melbourne, Victoria
- 3 Sites, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An expansion cohort of 20 subjects in Part 2 was originally planned to be recruited to study the optimum dose selected by the Steering Committee. However, the study was terminated at the end of Cohort 4 due to Sponsor decision in July 2019 and did not proceed to Part 2 of the protocol. The primary and secondary endpoints were analyzed based on data from the 24 subjects in Part 1.
Groups:
- Part 1: ASLAN003 100mg QD: ASLAN003: Patients will be administered with the study drug, ASLAN003. The study drug is to be administered orally, 100mg QD. Patients will receive a continuous 28-day treatment cycle of ASLAN003 at this dose until disease relapse, treatment failure (defined as failure to achieve a PR or higher within 4 cycles), development of unacceptable toxicity, withdrawal of consent or death. It is recommended to administer the study drug with food or within 30 minutes after food intake.
- Part 1: ASLAN003 200mg QD: ASLAN003: Patients will be administered with the study drug, ASLAN003. The study drug is to be administered orally, 200mg QD. Patients will receive a continuous 28-day treatment cycle of ASLAN003 at this dose until disease relapse, treatment failure (defined as failure to achieve a PR or higher within 4 cycles), development of unacceptable toxicity, withdrawal of consent or death. It is recommended to administer the study drug with food or within 30 minutes after food intake.
- Part 1: ASLAN003 100mg BID: ASLAN003: Patients will be administered with the study drug, ASLAN003. The study drug is to be administered orally, 100mg BID. Patients will receive a continuous 28-day treatment cycle of ASLAN003 at this dose until disease relapse, treatment failure (defined as failure to achieve a PR or higher within 4 cycles), development of unacceptable toxicity, withdrawal of consent or death. It is recommended to administer the study drug with food or within 30 minutes after food intake.
- Part 1: ASLAN003 200mg BID: ASLAN003: Patients will be administered with the study drug, ASLAN003. The study drug is to be administered orally, 200mg BID. Patients will receive a continuous 28-day treatment cycle of ASLAN003 at this dose until disease relapse, treatment failure (defined as failure to achieve a PR or higher within 4 cycles), development of unacceptable toxicity, withdrawal of consent or death. It is recommended to administer the study drug with food or within 30 minutes after food intake.
Period: Overall Study
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID
Started | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 1
Not completed — Disease recurrence | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 3 | 0 | 1
Not completed — Death | 1 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 2
Not completed — Disease progression (n=4), study closed by sponsor (n=1) | 3 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 0 | 2 | 8
  >=65 years | 2 | 4 | 6 | 4 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4 | 2 | 10
  Male | 2 | 6 | 2 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 5 | 5 | 4 | 15
  Asian | 5 | 1 | 1 | 1 | 8
  Other | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 24
Region of Enrollment [Number; unit: participants]
  Singapore | 4 | 1 | 1 | 1 | 7
  Australia | 2 | 5 | 5 | 5 | 17
Height [Mean (Standard Deviation); unit: CM] | 162.67 (8.189) | 173.25 (7.640) | 158.17 (9.827) | 164.17 (7.627) | 164.56 (9.604)
Weight [Mean (Standard Deviation); unit: KG] | 53.00 (13.549) | 82.32 (11.216) | 63.82 (16.551) | 81.72 (21.244) | 70.21 (9.637)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 19.855 (3.9883) | 27.368 (2.6446) | 25.065 (3.9042) | 30.553 (8.8254) | 25.710 (6.4119)

OUTCOME MEASURES:

1. Primary Outcome: Overall Complete Remission Rate
Description: Defined as the proportion of patients with a best response of complete remission (CR) or complete remission with incomplete hematologic recovery (CRi), defined in accordance with the IWG Response Criteria in AML from day 29. Treatment failure is defined as not achieving any response 4 months after study treatment. IWG Response Criteria in AML defines CR or CRi as:
  1. Complete remission (CR): Bone marrow blasts <5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions
  2. CR with incomplete recovery (CRi): All CR criteria except for residual neutropenia (<1.0 x 109/L (1000/µL)) or thrombocytopenia (<100 x 109/L (100,000/µL))
Time Frame: 4 months after study treatment
Population: The primary efficacy endpoint was OCRR, defined as the proportion of subjects with a best response of CR or CRi.
  The "Measure Type" and data in the "Outcome Measure Data Table" is reported as "Count of Participants" and corresponding proportion is provided next to the count.
  Two subjects who had major protocol deviations were excluded from the Evaluable for Response (EFR) analysis set. Primary and secondary efficacy analyses were performed on the EFR set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID
Number analyzed (Participants) | 6 | 4 | 6 | 6
Participants
  Responders | 0 | 0 | 0 | 0
  Treatment Failure | 2 | 4 | 2 | 6
  Non-evaluable | 4 | 0 | 4 | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events reported through 28 days post last study medication administration
Time Frame: Through 28 days post last study medication administration
Population: Overview of Treatment Emergent Adverse Events (TEAEs) - Safety Population
Measure: Number; unit: participants
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants
  Number of Patients with Any TEAE | 5 | 6 | 6 | 6
  Number of Patients with Any TEAE related to study treatment | 3 | 4 | 1 | 4
  Number of Patients with Any TEAE CTCAE grade 3 or higher | 5 | 5 | 6 | 6
  Number of Patients with Any TEAE CTCAE grade 3 or higher related to study treatment | 2 | 2 | 1 | 2
  Number of Patients with Any TEAE with outcome of death | 0 | 1 | 0 | 0
  Number of Patients with Any TEAE with outcome of death related to study treatment | 0 | 0 | 0 | 0
  Number of Patients with Any serious TEAE | 3 | 5 | 4 | 6
  Number of Patients with Any serious TEAE related to study treatment | 0 | 0 | 0 | 1
  Number of Patients with Any TEAE leading to discontinuation of study therapy | 0 | 0 | 1 | 0
  Number of Patients with Any TEAE leading to discontinuation of study therapy related to treatment | 0 | 0 | 0 | 0

3. Primary Outcome: Safety Assessments
Description: Safety Assessments - Clinical laboratory test: Hematology and Chemistry
Time Frame: Through 28 days post last study medication administration
Population: The Outcome Measure Data includes number of analyzed subjects who had abnormal values for hematology and chemistry parameters and reported as AEs by the Investigators. All 24 (100%) subjects enrolled in the study were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants
  Hematology - Abnormal white blood cell counts reported by Investigator as AEs of leukocytosis | 2 | 3 | 3 | 0
  Hematology - Abnormal/decreased hemoglobin values reported by Investigator as AEs of anaemia | 3 | 1 | 2 | 2
  Hematology - Abnormal neutrophil count reported by Investigator as AE of neutropenia | 0 | 0 | 0 | 1
  Hematology - Abnormal neutrophil counts reported by Investigator as AEs febrile neutropenia | 0 | 1 | 0 | 2
  Hematology - Abnormal/decreased platelet count reported by Investigator as AEs of thrombocytopenia | 2 | 0 | 2 | 1
  Chemistry - Abnormal serum potassium values reported by Investigator as AEs of hypokalaemia | 2 | 3 | 2 | 1
  Chemistry - Elevated levels of serum glucose reported by Investigator as AEs of hyperglycaemia | 1 | 1 | 0 | 0
  Chemistry - Abnormal blood creatinine reported by Investigator as AE of blood creatinine increased | 0 | 0 | 1 | 0

4. Secondary Outcome: Relapse Free Survival
Description: Defined as the time the criteria for remission (CR or CRi) are first met until there is evidence of patient relapse, regardless of whether the patient is still taking study drug. Relapse is defined as:
  * The reappearance of leukemic blasts in the peripheral blood or > 5% blasts in the bone marrow not attributable to any other cause;
  * The appearance of new dysplastic changes;
  * The reappearance of or development of cytologically proven extrameduallary disease;
  * The reappearance of a cytogenetic or molecular abnormality.
Time Frame: From 12 weeks post end of treatment (EOT) until the date of first documented relapse or date of death from any cause, whichever came first, assessed up to 24 months
Population: All the subjects were non-responders in this study, relapse free survival was not evaluated.
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Clinical Benefit Rate
Description: Defined as the proportion of subjects with an AML IWG best response of CR, CRi or PR. IWG Response Criteria in AML defines CR, CRi or PR as:
  1. Complete remission (CR): Bone marrow blasts <5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions
  2. CR with incomplete recovery (CRi): All CR criteria except for residual neutropenia (<1.0 x 109/L (1000/µL)) or thrombocytopenia (<100 x 109/L (100,000/µL))
  3. Partial remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5 to 25 percent; and decrease of pre-treatment bone marrow blast percentage by at least 50 percent
Time Frame: 4 months after study treatment
Population: In addition to achieving no responses (CR or CRi) for the primary endpoint, no PRs were achieved either, thus CBR was not evaluated.
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: % Change From Baseline in BM Blasts at Day 29
Description: Percent Change from Baseline in BM Blasts at Day 29
Time Frame: Baseline and day 29
Population: Only subjects with reduction of BM blasts evaluated on Day 29 are reported as % change from baseline in the Outcome Measure data.
Measure: Number; unit: Percentage change
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID
Number analyzed (Participants) | 1 | 1 | 0 | 0
Percentage change | -34.43 | -8.33 |  |

ADVERSE EVENTS:
Time Frame: From the time of informed consent and until 28 days after the last administration of study drug, up to 24 months.
Description: Definition of adverse event and/or serious adverse event, used to collect adverse event information, is the same with clinicaltrials.gov definition.
Arm/Group | Part 1: ASLAN003 100mg QD | Part 1: ASLAN003 200mg QD | Part 1: ASLAN003 100mg BID | Part 1: ASLAN003 200mg BID
All-Cause Mortality (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 3/6
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 4/6 | 6/6
Other Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 1/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: ASLAN003 100mg QD (N=6) | Part 1: ASLAN003 200mg QD (N=6) | Part 1: ASLAN003 100mg BID (N=6) | Part 1: ASLAN003 200mg BID (N=6)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathogen resistance (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: ASLAN003 100mg QD (N=6) | Part 1: ASLAN003 200mg QD (N=6) | Part 1: ASLAN003 100mg BID (N=6) | Part 1: ASLAN003 200mg BID (N=6)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (26)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT03451084/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03451084/SAP_003.pdf